CLINICAL TRIAL: NCT00161538
Title: A Randomized, Prospective Multicenter Study to Examine the Optimal Position of the Atrial Leads for Therapy of the Sinus Node Syndrome
Brief Title: Pacing of the Atria in Sick Sinus Syndrome Trial Preventive Strategies for Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic BRC (Industry)
Collaborators: Vitatron GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PASTA V.1.5
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2006-10-20 (Estimated); Status verified 2006-10

CONDITIONS: Sick Sinus Syndrome
Keywords: Cardiac Pacing, artificial; Atrial fibrillation; Pacemaker leads; Lead positions
MeSH Terms: conditions — Sick Sinus Syndrome; Atrial Fibrillation

INTERVENTIONS:
Device: Pacing leads to be implanted according randomization.
Device: Selection 9000 prevent AF an Diagnose AF

SUMMARY:
The purpose of this study is to determine which of 4 lead positions is most effective for pacemaker patients with Sick Sinus Syndrome in order to avoid development of atrial fibrillation.

DETAILED DESCRIPTION:
The incidence of Atrial Fibrillation (AF) in Sick Sinus Syndrome patients treated with pacing is quite high. As AF can cause dizziness, fatigue, thromboembolism and ischemic stroke it is clinically relevant. Due to earlier publications pacing modes and lead placement seem to influence the incidence of AF. In this study the incidence of AF will be compared between 4 different atrial lead positions:

1. Free atrial wall
2. right atrial appendage
3. coronary sinus-os
4. Dual site right atrial pacing: b) plus c).

The following primary parameters will be evaluated during the study period of 2 years after implantation:

1. Amounts of AF episodes with a duration of > 48 hours
2. Amounts of AF episodes with a duration of > 30 minutes
3. Consultations of physicians due to AF Secondarily, AF burden, Incidence of AF in total, Quality of Life, implant duration and complications will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Sick Sinus Syndrome
* Symptomatic sinus bradycardia
* Symptomatic SA block
* Bradycardia-Tachycardia-Syndrom
* Binodal diseases, Sinus Node Syndrome and high degree AV-Block
* In case of antiarrhythmic drug therapy: patient must be on a stable dose for at least 3 months before enrollment

Exclusion Criteria:

* Permanent atrial tachycardia that cannot be transferred into sinus rhythm by drugs or electric cardioversion
* Decompensated heart failure
* Dilatative cardiomyopathy with an ejection fraction < 35%
* Hypertrophic obstructive cardiomyopathy
* Symptomatic hypo- or hyperthyreosis
* Myocardial infarction less than 6 months ago
* Planned cardiac surgery intervention
* Pregnant woman
* Patients under 18 years of age
* Patients involved in other studies
* Patients, already implanted with other (cardiac) leads
* Patients with reduced expectancy of life due to other diseases
* Patients who are not able to agree in participation of the study
* Patients, who cannot attend follow-up visits due to their place of residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456
Dates: Start 2000-07; Study Completion 2006-06

PRIMARY OUTCOMES:
The incidence of AF is determined via memory of the pacemaker, which is saved at every follow-up visit at 1 and 10 days after implant and further on at 3, 6, 12, 18 and 24 months after implant.
24-Hour ECG and treadmill exercise as well as echocardiography shall be performed before implant and 6, 12 and 24 months after implant

SECONDARY OUTCOMES:
Treadmill exercise test as well as echocardiography shall be performed before implant and 6, 12 and 24 month after implant.
Quality of Life questionnaires are obtained before implant and 12 and 24 months after implants

CONTACTS AND LOCATIONS:
Overall Officials: Stefan G. Spitzer, MD, Principal Investigator
Locations (12):
- Germany (12):
  - Helios-Klinikum Aue, Aue
  - Klinikum Coburg, Coburg
  - Ambulantes Herz-Zentrum Dresden, Dresden
  - Werner-Forssmann-Krankenhaus GmbH, Eberswalde
  - Klinikum der Joh.-Wolfgang-Goethe-Universität, Frankfurt
  - Städtisches Krankenhaus Friedrichshafen, Friedrichshafen
  - Universitätskrankenhaus Eppendorf, Hamburg
  - Evang. Krankenhaus, Holzminden
  - Klinikum Ingolstadt, Ingolstadt
  - Evangelisches Krankenhaus Kalk GmbH, Köhl
  - Kreiskrankenhaus Leer, Leer
  - Krankenhaus Maria Hilf, Mönchengladbach

REFERENCES:
- [Background] Andersen HR, Nielsen JC, Thomsen PE, Thuesen L, Mortensen PT, Vesterlund T, Pedersen AK. Long-term follow-up of patients from a randomised trial of atrial versus ventricular pacing for sick-sinus syndrome. Lancet. 1997 Oct 25;350(9086):1210-6. doi: 10.1016/S0140-6736(97)03425-9. PMID 9652562
- [Background] Rosenqvist M, Brandt J, Schuller H. Long-term pacing in sinus node disease: effects of stimulation mode on cardiovascular morbidity and mortality. Am Heart J. 1988 Jul;116(1 Pt 1):16-22. doi: 10.1016/0002-8703(88)90244-x. PMID 3394616
- [Background] Prakash A, Saksena S, Hill M, Krol RB, Munsif AN, Giorgberidze I, Mathew P, Mehra R. Acute effects of dual-site right atrial pacing in patients with spontaneous and inducible atrial flutter and fibrillation. J Am Coll Cardiol. 1997 Apr;29(5):1007-14. doi: 10.1016/s0735-1097(97)00043-0. PMID 9120152